CLINICAL TRIAL: NCT02914743
Title: Providing Preventive Periodontal Treatment to Hospitalized Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Harvard School of Dental Medicine (Other)
Responsible Party: Principal Investigator, Matthew Tobey, Assistant in Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P001460
Record Dates: First submitted 2016-09-20; First posted 2016-09-26 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Type II Diabetes; Periodontal Disease
Keywords: Oral health; Diabetes; Interprofessionalism; Periodontal disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Periodontal Diseases; Diabetes Mellitus | interventions — Motivational Interviewing; Dental Prophylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dental Cleaning and MI Arm (Experimental): Subjects in this arm will receive a dental cleaning by the hygienist as well as a motivational interviewing (MI) session to explore the subject's motivations to pursue oral health treatment.
  Interventions: Behavioral: Motivational Interviewing; Procedure: Dental cleaning
- MI only Arm (Experimental): Subjects in this arm will not receive a dental cleaning but the hygienist will provide a motivational interviewing (MI) session to explore the subject's motivations to pursue oral health treatment.
  Interventions: Behavioral: Motivational Interviewing
- Control Arm (No Intervention): Subjects in this arm of the study will not receive any oral health intervention while hospitalized. A medical record review will be completed, and patients will be contacted via telephone at 3, 6, and 12 months post-hospitalization to assess their oral health-related quality of life and oral health care-seeking behaviors.

INTERVENTIONS:
Behavioral: Motivational Interviewing — This intervention will involve a discussion intended to explore subjects' motivations to pursue dental care and empower them to visit a dentist upon release from the hospital.
  Arms: Dental Cleaning and MI Arm; MI only Arm
Procedure: Dental cleaning — This procedure will involve the removal of plaque and supragingival and subgingival calculus from the surfaces of the teeth.
  Other Names: Dental prophylaxis
  Arms: Dental Cleaning and MI Arm

SUMMARY:
The purpose of this research intervention is to assess the oral health status and periodontal health of patients with diabetes hospitalized on a general medicine service, and to assess the effect of providing dental prophylaxis and motivational interviewing to patient health-seeking behaviors and provider attitudes towards oral health, as well as on patient health outcomes.

DETAILED DESCRIPTION:
Almost 20% of all patients admitted to the hospital carry a diagnosis of diabetes. Diabetes and periodontal disease have a bi-directional relationship; people with diabetes are at higher risk of tooth loss and poor oral health may impact nutrition and inflammation. Even among those with access to medical treatment for their diabetes, access to dental care may be challenging. In spite of their higher oral health risk, diabetic adults are less likely than their peers to attend a dental visit annually. While oral hygiene measures for ventilator-dependent patients have become standard of care, the oral health of less critically ill hospitalized patients has been noted to decline over the course of their hospitalization and patients generally do not have access to dental treatment., However, invasive dental treatment (restorations, tooth extraction, and periodontal scaling) has been demonstrated to be safe even for critically ill hospitalized patients. The inpatient setting, where patients are already receiving services from multiple disciplines and patients do not need to travel to see a healthcare provider, presents a unique opportunity to make integrative oral healthcare services accessible to diabetic patients, and to increase oral health knowledge of those health professionals caring for patients on an inpatient medical ward.

This study will involve provision of dental prophylaxis ("tooth cleaning") as well as motivational interviewing focused on oral health care-seeking behaviors provided by a dental hygienist to patients with a diagnosis of Type II diabetes who are hospitalized on a medicine floor of Massachusetts General Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patient has diagnosis of type 2 diabetes
* Patient has a primary care provider of record
* Patient is currently admitted to the house staff service of the Department of Medicine at MGH
* Patient is "ready or nearly ready for discharge," based on the assessment of the patient's medical team.

Exclusion Criteria:

1. History of cardiac conditions for which antibiotic prophylaxis is indicated prior to dental treatment per American Dental Association/American Heart Association guidelines:51

   1. Prosthetic cardiac valve or prosthetic material used for cardiac valve repair
   2. Previous infective endocarditis
   3. Congenital heart disease (CHD) encompassing:

   i. Unrepaired cyanotic CHD, including palliative shunts and conduits ii. Completely repaired congenital heart defect with prosthetic material or device, whether placed by surgery or by catheter intervention, during the first six months after the procedure iii. Repaired CHD with residual defects at the site or adjacent to the site of a prosthetic patch or prosthetic device (which inhibit endothelialization) d. Cardiac transplantation recipients who develop cardiac valvulopathy
2. Anticoagulated with International Normalized Ratio>2.5
3. History of prosthetic joint replacement in the last two years
4. Medical team declines enrollment
5. The patient is unable to participate in the provision of dental prophylaxis due to a medical condition such as altered mental status or altered cognitive status
6. Edentulous

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Dental care-seeking behavior | 12 months
  Subject-reported dental visit since hospitalization, assessed at 12 months after intervention.

SECONDARY OUTCOMES:
Healthcare costs | Up to 24 months
  Subject healthcare expenditures 12 months before and after intervention.
Oral health-related quality of life | 6 months
  Subject-reported oral health-related quality of life assessed at 6 months after intervention.
Change from baseline Hemoglobin A1c at 3 and 6 months | 6 months
  Subject Hemoglobin A1c reading as noted in electronic medical record 3 and 6 months after intervention.

OTHER OUTCOMES:
Clinician attitude towards the importance of oral health | 12 months
  Clinician attitudes towards the importance of oral health for patient wellbeing before and after working with the study's dental hygienist as measured by a Likert-scale question.
Clinician attitude towards the value of having a hygienist in the hospital setting | 12 months
  Clinician attitudes towards the value of working with a hygienist in the hospital setting before and after working with the study's dental hygienist as measured by a Likert-scale question.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Announcement of grant funding — http://hsdm.harvard.edu/news/dean%E2%80%99s-innovation-fund-recipients-announced